CLINICAL TRIAL: NCT04424030
Title: International Consortium for Multimodality Phenotyping in Adults With Non-compaction
Acronym: NONCOMPACT
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: The Cleveland Clinic (Other); University of Pennsylvania (Other); Erasmus Medical Center (Other); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Koen Nieman, Associate Professor of Medicine, Stanford University
Other Study IDs: 56001; SSU00099737 (Other: Advarra Single IRB)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Non-Compaction Cardiomyopathy
Keywords: Echocardiography; Magnetic resonance imaging; Computed tomography; Prognosis; Genetics
MeSH Terms: interventions — Echocardiography; Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After enrollment, blood will be drawn via venipuncture. The blood samples (35cc in total) will be centrifuged (15 minutes at 3500 RPM), after which the plasma, serum, red cells and buffy coat will be aliquoted from the vacutainers into color-coded vials. In addition to standard EDTA tubes we may include a CPT or PAX tube for more extensive analytics, or an Oragene tube for remote saliva collection. The aliquots and tubes will be stored at -70⁰C. The samples will remain at the site until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multimodality imaging: Patients who have undergone echocardiography and cardiac MRI as part of their clinical management A research cardiac CT scan will be performed in eligible participants
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Computed tomography (CT)

INTERVENTIONS:
Diagnostic Test: Echocardiography — Standard echocardiography exam performed as part of clinical management.
Diagnostic Test: Magnetic resonance imaging (MRI) — Standard comprehensive cardiac MRI exam of the heart performed as part of clinical management.
Diagnostic Test: Computed tomography (CT) — ECG-triggered, contrast-enhanced CT scan of the heart performed for research purposes in eligible study participants.

SUMMARY:
Non-compaction cardiomyopathy (NCCM) is a heterogeneous, poorly understood disorder characterized by a prominent inner layer of loose myocardial tissue, and associated with heart failure, stroke, severe rhythm irregularities and death. For a growing population diagnosed with NCCM there is a need for better risk stratification to appropriately allocate (or safely withhold) these impactful preventive measures. The goal of this international consortium is to improve care of patients with non-compaction cardiomyopathy. We hypothesize that comprehensive analysis of clinical, genetic, structural and functional information will improve risk stratification. In addition, we hypothesize that detailed structural analysis will allow for differentiation of pathological and benign patterns of non-compaction. In a large cohort of adult patients with suspected NCCM we will perform in-depth phenotyping, including clinical information, pedigree data, genetics, echocardiography and MRI, and follow patients for up to 3 years. We will apply machine-learning based analytics to develop predictive models and compare their performance to currently used models and treatment criteria. Secondly, in a subset of patients we will perform high-resolution cardiac CT for detailed structural characterization of the myocardial wall. We will investigate associations between myocardial structure and regional contractile function, as assessed by echo and MRI. The aim of this proposal is to identify a structural signature associated with pathological non-compaction and improve developed risk prediction models. Discovery of pathological structural signatures through innovative imaging techniques, in relation to myocardial contractility, will advance our understanding of NCCM.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Hypertrabeculation of the left ventricle fulfilling the echo-based Jenni criteria of NCCM
* Clinical cardiac MRI examination performed or planned

Exclusion Criteria (general cohort):

* Complex congenital disease (including transposition great arteries, tetralogy of Fallot, tricuspid atresia, truncus arteriosis, single ventricle, hypoplastic left heart, pulmonary atresia, double-outlet RV), neuromuscular disorders or isolated RV non-compaction
* Inability to provide informed consent
* Contra-indications to MRI, which apply if the clinical cardiac MRI has not yet been performed at the time of study enrollment: permanent pacemakers/ICDs, MRI contrast medium allergy, significant arrhythmia with highly irregular RR intervals, severe dyspnea with inability to lay flat/breath hold, inability to communicate with the MRI technician or follow commands for any reason (psychosis, agitation, etc.), other site-specific contra-indications to clinical MRI of the heart.

Exclusion Criteria (cardiac CT examination):

* Age <21 years
* Decompensated heart failure, or otherwise clinically unstable
* BMI>40 kg/m2
* Pregnancy (or cannot be ruled out)
* Known iodine contrast medium allergy
* Kidney dysfunction: eGFR<45 ml/min
* Thyroid disease: toxic multinodular goiter, Graves' disease, Hashimoto's thyroiditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertrabeculation of the left ventricle fulfilling echo-based criteria of non-compaction cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hard embolic adverse events | Up to 4 years after enrollment
  Clinical neuro/systemic embolic event by autopsy, imaging or specialist evaluation
Incidence of hard arrhythmic adverse events | Up to 4 years after enrollment
  Sudden death (aborted), appropriate ICD discharge or VT/VF on ECG or rhythm/device monitoring

SECONDARY OUTCOMES:
Incidence of hard heart failure related adverse events | Up to 4 years after enrollment
  Heart failure death, cardiac transplantation or mechanical circulatory support
Incidence of composite of hard adverse events | Up to 4 years after enrollment
  Hard embolic, arrhythmic and heart failure related adverse events (as described above)
Incidence of all embolic adverse events | Up to 4 years after enrollment
  Hard embolic adverse events or transient neurologic event without objective infarction
Incidence of all arrhythmic adverse events | Up to 4 years after enrollment
  Hard arrhythmic adverse events or syncope without recorded arrhythmia
Incidence of all heart failure related adverse events | Up to 4 years after enrollment
  Hard heart failure related adverse events or resynchronization therapy, heart failure hospital admission
Incidence of composite of adverse events | Up to 4 years after enrollment
  All embolic, arrhythmic or heart failure related adverse events (as described above)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD, PhD, Principal Investigator — Stanford University
Locations (5):
- United States (3):
  - Stanford University, Palo Alto, California
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Erasmus Medical Center, Rotterdam, Netherlands
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be created and maintained on a public website in a password-protected area, where the frequency of use of the datasets can be monitored by Stanford and NHLBI.